CLINICAL TRIAL: NCT04423705
Title: The Turkish Version of The Active-Q: Physical Activity Questionnaire: A Reliability and Validity Study
Brief Title: The Turkish Version of The Active-Q: Physical Activity Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Pınar Kısacık, PhD, Principle Investigator, Hacettepe University
Other Study IDs: GO 19/776
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Exercise; Validity; Reliability
Keywords: The Active-Q Scale; Physical activity; Validation studies; Turkish
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators think that "The Active-Q: Physical Activity Questionnaire" will help physiotherapists and other health professionals in the field and in the field to evaluate individuals' physical activity by revealing their energy consumption values. Therefore, it was aimed to make this scale available to Turkish healthcare professionals by conducting the Turkish validity and reliability study.

DETAILED DESCRIPTION:
Individuals forming modern societies along with technological developments are increasingly adopting sedentary lifestyle. This situation increases the risks in terms of morbidity and mortality. For this reason, especially all countries build their health policies on increasing physical activity and make strides to improve it. In order to reach the ideal physical activity level, the physical activity level should be evaluated. However, when the literature is evaluated, it is possible to come across different and many physical activity evaluation methods. This makes it difficult to compare. On the other hand, many researchers prefer to use scales and surveys because of their low costs and ease of use. Although there are many physical activity assessment scales in the literature based on age, gender, disorder or disease, social needs and other features, many of them cannot be used in our society because they are not Turkish. This poses an important obstacle for Turkish researchers to evaluate physical activity.

"The Active-Q: Physical Activity Questionnaire" is a web-based scale developed to investigate the absence of physical activity and activity for individuals over the age of 18. Individuals are asked to answer questions about their activity habits in the past year. By developing the scale, Bonn et al. Tested its validity and reliability comparatively with the 'Double labeled water' method and the accelerometer.

The investigators think that "The Active-Q: Physical Activity Questionnaire" will help physiotherapists and other health professionals in the field and in the field to evaluate individuals' physical activity by revealing their energy consumption values. Therefore, it was aimed to make this scale available to Turkish healthcare professionals by conducting the Turkish validity and reliability study.

ELIGIBILITY:
Inclusion Criteria:

* to be a native Turkish speaker
* to be a volunteer

Exclusion Criteria:

* to make any form of weight alternation diet
* to be pregnant
* to have given birth during last 1 year
* to have any chronic and/or orthopedic disease/problem/syndrome
* to have any traumatic injury or any form of surgery during last 1 year

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants of both sexes, aged 20 to 65 years recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Reliability: The Active-Q | 2 months
  To measure stability of the test over time by The Active-Q: Physical Activity Questionnaire. The Active-Q is filled with one week interval.
Validity- IPAQ-SF | 2 months
  To test in order to establish the correlation among the proposed instrument and instruments that had already been translated and validated. The Short Form of the International Physical Activity Questionnaire (IPAQ-SF) is used.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Karagül, Mac, Principal Investigator — Hacettepe University; Sibel Bozgeyik, PhD, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: No